CLINICAL TRIAL: NCT03355040
Title: Induction of Labour for LGA fœtus in Women Without Insulin-treated Diabetes.. Application of DAME Study in Montpellier University Hospital.
Brief Title: Induction of Labour for LGA fœtus in Women Without Insulin-treated Diabetes.
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0261
Record Dates: First submitted 2017-10-12; First posted 2017-11-28 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Macrosomia; Induction of Labour; Non-insulin-dependent Diabetes
Keywords: shoulder dystocia; maternal and neonatal morbidity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Shoulder Dystocia | interventions — Labor, Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: induction of labour — induction of labour

SUMMARY:
A french study published in 2015 (DAME) showed a decrease of shoulder dystocia and an increase of spontaneous vaginal delivery when the non insulin-treated diabetes patients with large-for-date fetus were induced.

This new protocole was introduced in Montpellier University Hospital delivery room.

The aim of this study is to evaluate the protocole in Montpellier hospital and to compare our results with the DAME results.

DETAILED DESCRIPTION:
Currently, large for date fœtus need an induction of labour just if the mother is an insulin diabetic.

The DAME's protocol included the large for date feotus witch have a estimate weight >3500g at 36 GA, >3700g at 37 GA, >3900g at 38 GA.

ELIGIBILITY:
Inclusion criteria:

Age >18 years old Single pregnancy Cephalic presentation no contraindications to planned vaginal delivery no fœtal pathology

Large-for-date foetus (estimated weight > 95%) :

* Clinically suspeted or estilated weight >90% at the 3 trimester ultrasound
* Estimated fœtal weight :

> 3500g at 36 GA > 3700g at 37 GA > 3900g at 38 GA

Exclusion criteria:

Age <18 yeaurs old contraindications to vaginal delivery insulin-trated diabetics or imbalance diabetics. neonatal trauma or shoulder dystocia, severe urinary or faecal incontinence.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant patients non diabetic or diabetic without insulin-treatment with large for date fœtus.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
number of shoulder dystocia | 1 day (after delivery)
  number of shoulder dystocia
number of Clavicle fracture | 1 day (after delivery)
  number of Clavicle fracture
number of Brachial plexus injury | 1 day (after delivery)
  number of Brachial plexus injury
number of Intracranial heamorrhage | 1 day (after delivery)
  number of Intracranial heamorrhage
number of Neonatal death | 1 day (after delivery)
  number of Neonatal death

SECONDARY OUTCOMES:
Number of Cord blood pH< 7,10 for the newborn | 1 day (after delivery)
  Number of Cord blood pH< 7,10 for the newborn
Number of apgar < 7 at 5 min for the newborn | 1 day (after delivery)
  Number of apgar < 7 at 5 min for the newborn
Number of admission to neonatal intensive care unit for the newborn | 1 day (after delivery)
  Number of admission to neonatal intensive care unit for the newborn
Number of highest bilirubin concentration for the newborn | 1 day (after delivery)
  Number of highest bilirubin concentration for the newborn
Number of Caesarean for the patient | 1 day (after delivery)
  Number of Caesarean for the patient
Number of Forceps or vacuum for the patient | 1 day (after delivery)
  Number of Forceps or vacuum for the patient
Number of Haemorrage and blood transfusion for the patient | 1 day (after delivery)
  Number of Haemorrage and blood transfusion for the patient
Number of Anal sphincter tear for the patient | 1 day (after delivery)
  Number of Anal sphincter tear for the patient

CONTACTS AND LOCATIONS:
Overall Officials: florent FUCHS, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC